CLINICAL TRIAL: NCT03954080
Title: Trialing of Intra-spinal Stimulation in Patients With Complex Regional Pain Syndrome or Causalgia
Brief Title: Trialing of ISS in Patients With CRPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Millennium Pain Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-2019ISS/CRPS
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: CRPS I; Causalgia
MeSH Terms: conditions — Causalgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ISS (Experimental)
  Interventions: Device: Intraspinal-optimal stim therapy

INTERVENTIONS:
Device: Intraspinal-optimal stim therapy — During the trial, percutaneous lead(s) will be implanted, following standard clinical practices, in the posterior epidural space with the final lead position located in the optimal area to provide pain relief by stimulating neural tissue in order to create paresthesia(s) only on the painful dermatome(s). During Intraspinal-Optimal Stim, a set of electrodes in the stimulation lead(s) will deliver a charge-balanced, pulsed electrical signal with stimulation parameters (frequency, pulse width, and amplitude) within the FDA approved specifications of the commercially available external neurostimulator. These will be adjusted to produce paresthesia coverage of the painful area. Patients that will report equal or greater than 50% reduction in pain, relative to baseline pain, may undergo permanent implantation of a commercially available neurostimulator (INS). This will require a surgical intervention to implant stimulation leads, INS and anchoring hardware followed by therapy programming.

SUMMARY:
This is a multi-center, prospective, open-label, single-arm, observational, feasibility study. The goal of this study is to determine the feasibility of intra-spinal stimulation with optimal paresthesia coverage therapy for chronic pain relief in patients with complex regional pain syndrome type I or causalgia. Up to 20 patients with intractable chronic severe limb pain associated with complex regional pain syndrome (CRPS) will be included in the study. A standard of care trial phase to test a subjects' response to Intraspinal-Optimal Stim therapy will be conducted during a 3 to 10-day period. Patients that obtain 50% or greater pain relief during the trial period will undergo permanent implantation of the device. Primary outcome will evaluate pain response at 3 months of therapy, based on NPRS pain score relative to baseline. Patients will be followed up for 6 months after the start of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent to participate in this clinical study.
2. Must be 18 years old or older.
3. Predominant pain in one or both of the lower limbs attributed to CRPS or causalgia that has been refractory to conservative therapy for at least 3 months.
4. Average pain intensity larger or equal to 6 on the numeric pain rating scale (NPRS).
5. Appropriate candidate for spinal cord stimulation as determined by the Investigator.
6. Subjects must be on a stable dose of pain medication regimen for at least 1 month.
7. Must be able to comply with the requirements of study visits.
8. Have cognitive ability of operate the remote control and follow therapy instructions and directions by clinicians.

Exclusion Criteria:

1. Systemic infection.
2. Any other active implanted device.
3. Evidence of serious neurological, psychological or psychiatric disorders.
4. Previous posterior decompressive laminectomy that precludes appropriate posterior epidural placement of stimulation lead(s).
5. Patient who are pregnant, breast-feeding or women of childbearing potential with positive pregnancy tests.
6. Human immunodeficiency virus (HIV) infection or a clinically significant infection.
7. A clinically significant disorder such as cerebrovascular disease, pulmonary infarction, ischemic heart disease, cardiac dysrhythmia, myocardial infarction, or congestive heart failure or any other as determined by the investigator.
8. Uncontrolled diabetes, uncontrolled pulmonary disease, or uncontrolled hypertension.
9. Patients who have evidence of major psychiatric disease, mental disorder, drug dependency, alcohol dependency, or substance abuse disorders.
10. Patients who have progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, acute herniated disc, or any other as determined by investigator.
11. Medical condition or pain in other body areas determined by the Investigator as interfering with study procedures, accurate pain reporting, and/or confound evaluation of study end points.
12. Concurrent participation in another clinical study.
13. Involvement in an injury or disability claim under current litigation or a pending or approved workers' compensation claim.
14. Escalating or changing pain condition over the last 30 days that creates difficulty of pain evaluation by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in pain relative to baseline pain (i.e. prior to therapy) at 3 months after device activation for providing Intraspinal-Optimal Stim therapy | 3 months after therapy activation
  Change in pain relative to baseline pain (i.e. prior to therapy) at 3 months after device activation for providing Intraspinal-Optimal Stim therapy. Pain scoring will be based on the 11-points (0 to 10) numerical pain rating scale. In this scale a value of 0 means no pain, and a value of 10 reflects the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Vallejo, MD,PhD, Principal Investigator — Millennium Pain Center
Locations (1):
- Millennium Pain Center, Bloomington, Illinois, United States

REFERENCES:
- [Derived] Vallejo R, Fishman MA, Shah B, Kim P, Benyamin R, Vetri F, Tilley DM, Cedeno DL. Targeted Nerve Root Stimulation Alleviates Intractable Chronic Limb Pain Associated with Complex Regional Pain Syndrome - A Prospective Multi-Center Feasibility Study. Pain Physician. 2024 May;27(4):213-222. PMID 38805527